CLINICAL TRIAL: NCT05637918
Title: The Relationship Between Gastric Ultrasound Findings and Endoscopically Aspirated Volume in Infants and Determination of Antral Cut-off Value for the Diagnosis of Empty Stomach
Brief Title: Ultrasound for Prediction of Empty Stomach in Infants
Status: Completed | Type: Observational
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Feyza Sever, Principal investigator, Ankara City Hospital Bilkent
Other Study IDs: E2-21-490
Record Dates: First submitted 2022-11-24; First posted 2022-12-06 (Actual); Last update posted 2022-12-14 (Actual); Status verified 2022-11

CONDITIONS: Children, Only; Pulmonary Aspiration; Anesthesia; Fasting
Keywords: Gastric ultrasound; Infant; Upper gastrointestinal endoscopy; Empty stomach
MeSH Terms: conditions — Fasting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1 (Patients who recorded as Grade 0): Patients whose antrum appears empty in supine and right lateral decubitus (RLD) positions by gastric ultrasound (Grade 0). Groups are classified according to the qualitative evaluation of the antrum by gastric sonographic examination.
  The nature of the gastric contents (empty, clear liquid, dark liquid/solid) is established based on the qualitative findings by gastric antral ultrasonography. The qualitative evaluation of the antrum was recorded according to the 3-point grading system as Grade 0, Grade 1, and Grade 2.
  Grade 0: antrum appears empty in both positions. Grade 1: antrum appears empty in the supine position but a small volume of gastric clear fluid is visible in the RLD position.
  Grade 2: antral clear fluid visualized in both the supine and RLD position
  Interventions: Other: Group 1 (Patients who recorded as Grade 0)
- Group 2 ( Patients who recorded as Grade 1): Patients whose antrum appears empty in the supine position but a small volume of gastric clear fluid is visible in the RLD position by gastric ultrasound (Grade 1). Groups are classified according to the qualitative evaluation of the antrum by gastric sonographic examination The nature of the gastric contents (empty, clear liquid, dark liquid/solid) is established based on the qualitative findings by gastric antral ultrasonography. The qualitative evaluation of the antrum was recorded according to the 3-point grading system as Grade 0, Grade 1, and Grade 2.
  Grade 0: antrum appears empty in both positions. Grade 1: antrum appears empty in the supine position but a small volume of gastric clear fluid is visible in the RLD position.
  Grade 2: antral clear fluid visualized in both the supine and RLD position
  Interventions: Other: Group 2 ( Patients who recorded as Grade 1)

INTERVENTIONS:
Other: Group 1 (Patients who recorded as Grade 0) — When the gastric contents were evaluated with the upper gastrointestinal endoscopy, the stomach was completely empty in Group 1 that patients who recorded as Grade 0.
  Groups: Group 1 (Patients who recorded as Grade 0)
Other: Group 2 ( Patients who recorded as Grade 1) — When the gastric contents were evaluated with the endoscope, small volume of gastric clear fluid was visible and gastric content aspirated and measured in Group 2 that patients who recorded as Grade 1.
  Groups: Group 2 ( Patients who recorded as Grade 1)

SUMMARY:
Background and Aim: Pulmonary aspiration of gastric content is a serious perioperative complication. What is known about the pediatric patient's fasting time is usually based on parental history alone, but in some situation there may be doubts about an empty stomach in young children. Ultrasound examination of the gastric antrum is increasingly used and is emerging as a valuable perioperative noninvasive tool for the indirect assessment of gastric volumes in children. The objective of this prospective study was to assess the relationship between the cross-sectional area (CSA) of the antrum measured by gastric ultrasound and gastric volumes suctioned endoscopically, also to determine the best cut-off value of CSA for empty antrum in the pediatric population less than 24 months of age.

DETAILED DESCRIPTION:
Protocol: This study was performed in Pediatric Gastrointestinal (GI) Endoscopy Unit after receiving Institutional Ethics Board approval. Following induction of anaesthesia, antral sonography was performed in supine and right lateral decubitus (RLD) positions in 46 fasted infants prior to upper GI endoscopic evaluation. Antral CSA measurements in both positions and the qualitative evaluation of the antrum (according to the 3-point grading system) were recorded. Grade 0: antrum appears empty in both positions. Grade 1: antrum appears empty in the supine position but a small volume of gastric clear fluid is visible in the RLD. Grade 2: antral clear fluid visualized in both the supine and RLD position. The calculation of the antral CSA was performed by measuring the longitudinal diameter (D1) and the antero-posterior diameter (D2) of the antrum at rest, between peristaltic contractions, from serosa to serosa. Cross-sectional area was calculated using the standard formula for surface area of an ellipse CSA= π x D1 x D2 / 4. Gastric contents were endoscopically suctioned and measured by a graduated specimen trap with 1 ml increments.

Sample size A sample of 23 from the positive group and 23 from the negative group achieve 80% power to detect a difference of 0,2300 between the area under the receiver operating characteristic (ROC) curve (AUC) under the null hypothesis of ,5000 and an AUC under the alternative hypothesis of 0,7300 using a two-sided z-test at a significance level of 0,05000. The data are continuous responses. The AUC is computed between false positive rates of 0,000 and 1,000. The ratio of the standard deviation of the responses in the negative group to the standard deviation of the responses in the positive group is 1,000.

Statistical analysis:

All statistical analysis was performed using IBM SPSS for Windows Version 23.0 software. Descriptive statistics for continuous variables were shown as mean ± standard deviation (SD) or median [inter-quartile range (IQR); 25-75th percentile]. Categorical variables were shown as the number of patients and percentage (%). Whether the distributions of continuous variables were normal or not was determined by the Shapiro Wilks test. Correlations between continuous variables were given by Spearman Correlation Coefficient. Discriminative ability of the CSA was determined by ROC curve analysis. Optimal cut-off value was given by Youden index. Sensitivity, specificity, positive and negative predictive value were calculated at this point. A p value less than 0.05 was considered statistically significant.

Stepwise linear regression analysis was applied to estimate CSA. The variables those p values <0.20 in the univariate analysis were included in multiple regression model. The independent variables were determined as age, BMI and CSA-RLD. The adequacy of the established regression models was demonstrated by R2.

ELIGIBILITY:
Inclusion Criteria:

* All infants (< 24 months age) undergoing elective upper GI endoscopy under general anesthesia and American Society of Anesthesiology (ASA) physical status I -II, were included in this study

Exclusion Criteria:

* Parental refusal
* Previous lower esophageal or gastric surgery
* Non-adherence with the fasting regimen
* More than 5 minutes between gastric sonography and endoscopy

Max Age: 24 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Infants (< 24 months age) undergoing elective upper GI endoscopy
Sampling Method: Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
The relationship between antral cross-sectional area and aspirated gastric volumes | 30 minutes
  The investigators wanted to evaluate the correlation between sonographically measured gastric antral CSA in both supine and RLD positions, and gastric volume suctioned under direct endoscopic visualization in infants between 0-24 months age.
The best cut-off value of CSA for an empty antrum | 30 minutes
  The investigators wanted to determine the best cut-off value of CSA for a truly empty antrum in the pediatric population less than 24 months of age

SECONDARY OUTCOMES:
A mathematical model for gastric volume estimation | 30 minutes
  The investigators wanted to generate a final predictive model for gastric volume estimation in infants.

CONTACTS AND LOCATIONS:
Overall Officials: Feyza Sever, Principal Investigator — Ankara City Hospital Bilkent
Locations (1):
- Feyza Sever, Ankara, Çankaya, Turkey (Türkiye)